CLINICAL TRIAL: NCT06219395
Title: Diagnostic Yield of Video Capsule Endoscopy for Iron Deficiency Anaemia
Brief Title: Capsule Endoscopy in Iron Deficiency Anaemia
Acronym: WCE-IDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 281233
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Iron Deficiency Anemia; Bowel Cancer
MeSH Terms: conditions — Anemia, Iron-Deficiency; Intestinal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Iron deficiency anaemia: Persons 18-85 years with Iron deficiency anaemia referred for gastroscopy and colonoscopy
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Patients will be examined with gastroscopy, colonoscopy and WCE and the diagnostic yield of combined gastroscopy/colonoscopy will be compared to WCE

SUMMARY:
This project aim to investigate whether wireless capsule endoscopy(WCE) has a similar diagnostic yield as conventional endoscopy in detecting the cause of iron deficiency anemia (IDA)

DETAILED DESCRIPTION:
IDA is common and 90-95% of cases are caused by bleeding from ulcers, tumours or vascular malformations in the oesophagus, stomach, duodenum, small intestine or the large bowel.Bleeding from more than one localisation is common.

International guidelines recommend bidirectional endoscopy(gastro- and colonoscopy) to detect and treat the source of bleeding.

Our hypothesis is that WCE is non-inferior to the combination of gastroscopy and colonoscopy in locating GI-bleeding and that complete examinations will be achieved in ≥90% of the examinations.

ELIGIBILITY:
Inclusion Criteria:

* Referred to flexible endoscopy for a verified Iron Deficiency Anaemia

Exclusion Criteria:

* Unwillingness to participate
* Not able to provide informed consent
* Not understanding the instructions
* Severe cardio-vascular disease New York Heart Association III-IV
* Symptoms of bowel obstruction/previous bowel obstruction
* Bowel surgery except for end to end anastomosis in the colon
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons with Iron Deficiency Anaemia referred for endoscopic diagnostic work-up
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 90 minutes
  Mucosal lesions detected

SECONDARY OUTCOMES:
Small bowel lesions | 90 minutes
  Number of lesions detected in the small bowel
Complete examination | 90 minutes
  Proportion of complete examinations
Bowel preparation | 90 minute
  Proportion of satisfactory bowel preparation
Adequate examinations | 90 minutes
  Proportion of adequate examinations defined as both satisfactory bowel preparation and complete examination

CONTACTS AND LOCATIONS:
Overall Officials: Thomas de Lange, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided